CLINICAL TRIAL: NCT03211325
Title: Identification of Transient Receptor Potential (TRP) Channels as New Potential Therapeutic Targets in Primary and Secondary Raynaud's Phenomenon.
Brief Title: Identification of TRP Channels as New Potential Therapeutic Targets in Primary and Secondary Raynaud's Phenomenon.
Acronym: TRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC15.164
Record Dates: First submitted 2017-06-20; First posted 2017-07-07 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2019-04

CONDITIONS: Raynaud's Phenomenon Isolated Primary; Raynaud's Phenomenon (Secondary); Healthy
Keywords: Transient Receptor Potential Channels; Raynaud's Phenomenon Isolated Primary; Raynaud's Phenomenon (Secondary)
MeSH Terms: conditions — Raynaud Disease | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy (Experimental): Two sequences of ten healthy volunteers each will be performed :
  During the first sequence, a biopsy of the gluteal area and another of the surrounding nail area of a finger will be sampled.Then, the cutaneous blood flux of the hand will be recorded at rest and during cooling and warming periods.
  During the second sequence, two other biopsies of the surrounding nail area of two other fingers will be sampled.
  Interventions: Procedure: Biopsy
- Primary Raynaud's phenomenon (Experimental): Two sequences of ten primary Raynaud's syndrome each will be performed :
  During the first sequence, a biopsy of the gluteal area and another of the surrounding nail area of a finger will be sampled.Then, the cutaneous blood flux of the hand will be recorded at rest and during cooling and warming periods.
  During the second sequence, two other biopsies of the surrounding nail area of two other fingers will be sampled.
  Interventions: Procedure: Biopsy
- Secondary Raynaud's phenomenon (Experimental): Two sequences of ten patients each will be performed :
  During the first sequence, a biopsy of the gluteal area and another of the surrounding nail area of a finger will be sampled.Then, the cutaneous blood flux of the hand will be recorded at rest and during cooling and warming periods.
  During the second sequence, two other biopsies of the surrounding nail area of two other fingers will be sampled.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy

SUMMARY:
The investigators seek to perform a comparative transcriptome analysis of TRP channels residing in the skin between primary and scleroderma secondary Raynaud's phenomenon and healthy subjects.

DETAILED DESCRIPTION:
Raynaud's phenomenon (RP) is a clinical syndrome that results from an excessive vascular reactivity of the microcirculation of the fingers and/or other extremities of the body in response to a stress, mostly cold.

Primary RP affects 4 to 6% of the general population and displays important geographic variations. Most secondary RP are linked to systemic scleroderma, a rare condition affecting mainly women. The systemic scleroderma is characterized by a cutaneous and visceral fibrosis and is associated with micro vascular damages and the production of self antibodies directed against specific cellular antigenes. The American College of Rheumatology in association with the European League Against Rheumatism has recently set diagnostic criteria that define this disease more precisely. Besides, clinical forms without cutaneous infringment have been described as limited scleroderma. Cutaneous limited forms are characterized by cutaneous fibrosis affecting mainly hands, arms and face.

RP is the first clinical sign of these forms ; anti-centromer antibodies are found in 50 to 90% patients. Diffuse cutaneous scleroderma is a fast progressing disease that affects most parts of the skin and internal organs and displays the presence of anti topoisomerase antibodies in 30% of the patients.

Whether it is primary or secondary, severe forms of RP can result in an important functional disability. Besides that, iterative ischemic episodes contribute to the onset of trophic disorders that are associated with a higher morbidity. These trophic disorders are mainly encountered in the most severe forms, especially those that are secondary to systemic scleroderma ; a third of which will turn into gangrene or amputation, leading to an important disability for these patients. Up to now, no curative treatment of these ulcers has displayed a convincing efficacy.

Despite its frequency and the potential seriousness of its complications, therapeutic care options for RP remain limited. Conservative measures are recommended in the first place, especially avoiding cold exposure and wearing warm clothes. When those measures do not suffice, pharmacological treatment can be introduced. Only calcic inhibitors are authorized for this indication but their effect on the frequency of the crises is modest (reduction of 2.8 crises per week on average). In scleroderma secondary RP, the effect appears to be modest as well according to the severity of the affection and displays a reduction of 4 crises per week on average. Besides that, this kind of treatment, when taken continuously, exposes the patients to side effects (inferior limb edema in particular). Other vasodilators such as type 5 phosphodiesterase have a significant effect, but the latter remains low in secondary RPs. Finally, intravenous injections of Iloprost on a sequential scheme have displayed a superior effect compared to Nifedipine, but result in intense and frequent side effects that limit considerably the use of this medication for a common practice.

Therefore, there is a real need for new therapeutic targets in RP and this requires a better knowledge of the physiopathology of this phenomenon.

Whether it is primary or secondary, microvascular dysfunction is now considered as a key element in the physiopathogeny of RP. Some ionic channels from the Transient Receptor Potential Channels' family react to temperature variations and are therefore involved in the microvascular response. In the cutaneous tissue, multiple TRP channels are present on the afferent neurons and are involved in the response to hot temperatures (especially TRPV1, TRPV3 and TRPV4) or to environmental cold (TRPM8) or hyper algic cold (TRPA1). Although they were initially reduced to an afferent role towards thermic or chemical stimuli, TRP channels have been lately recognized as having more complex functions, especially in the cutaneous homeostasis sustainibility, the growth and cellular differentiation and even the inflammatory response. Thus, the recent identification of numerous TRP channels (TRPV1, TRPV3, TRPV4, TRPM8, TRPA1, TRPC1, TRPC4, TRPV6) on the surface of keratinocytes suggests their involvement in the differenciation of these cells. Although their precise role and barrier function in the skin remain unknown, anomalies of the expression of some TRP channels have been associated with specific dermatologic diseases, and have recently being the issue of a review. Nevertheless, TRP expression in Raynaud's phenomenon has been investigated only few times in human skin .

Considering the major role of the micro vascular dysfunction in RP and the involvement of specific TRP channels in the regulation of the cutaneous microvascular tone, the investigators put forward the hypothesis that the expression of some of these channels could be modified in primary and scleroderma secondary RP forms. This hypothesis is supported by an experimental trial (on mouse model of systemic cutaneous scleroderma), in which the activation of TRPV1 has been associated to the release of vasodilator peptides that displayed a protective effect against fibrosis and thus suggesting a plausible role of TRPV1 in the physiopathology of cutaneous systemic scleroderma.

Although RP strikes different parts of the body (hands, feet, ears...), the essential topography of Raynaud's crises remains hands. In scleroderma secondary RP, the microcirculatory damages that are the easiest to reach are the areas surrounding nails. The latters can be examined using a non-invasive technique that is capillaroscopy and sometimes even to the naked eye. Histology by cutaneous biopsy can be made as well.

The investigators propose here to sample cutaneous biopsies in these areas, that are on the one hand the most pathognomonic to display the microvascular damages and on the other hand, concerned by the Raynaud's crises.

Now studied as potential therapeutic targets for many disorders, TRP channels could represent a very interesting track in severe RP forms. The current development of numerous agonists and inhibitors of TRP channels could allow to foresee a clinical trial in Raynaud's phenomenon. On a physiopathological point of view, a better knowledge of the potential role of TRP channels in this disease could also explain the differences that have been observed between primary and secondary Raynaud's phenomenons.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers :dated and signed written consent
* Primary Raynaud's patients :
* dated and signed written consent
* subject presenting a primary Raynaud's phenomenon non associated to a connectivite. RP crisis are defined by a succession of caracteristic symptoms : a syncopal phase with distal whitening of the fingers, usually followed by a cyanotic phase, and then a hyperhemic phase with the outbreak of painful redness.The syncopal phase is always present, while the two other phases can be less pronounced, or even absent.
* Sclerodermy secondary Raynaud's patients :
* dated and signed written consent
* subject with Raynaud's phenomenon secondary to systemic sclerosis, according to the 2013 EULAR/ACR criteria.

Exclusion Criteria:

* Minor person or major person protected by the law
* Exclusion period for any clinical trial including a medication or focusing on a clinical device linked to the pathology
* Social secutrity scheme non-affiliated person or person who cannot pretend to such a scheme
* Pregnant woman, parturient or breast-feeding mother
* Person displaying a digital ulcer or a history of digital ulcer
* Severe concurrent disease found at oral questioning : evolutive cancer, hepatic insufficiency, history of myocardic infarction in the past five years, angina pectoris
* Hemodynamic instability
* Any tobacco consumption
* Any contraindication to the medication used in this trial :
* Anesderm ® (lidocain/procain) : Known hypersensitivity, to local amide linking anesthetic or to any other compound of the cream, congenital methemoglobin porphyria
* Lidocain Aguettant 5 mg/ml without preservative, injectable solution : Known hypersensitivity to lidocain chlorhydrate, to local amide linking anesthetic or to one of its excipients, patients affected with reccurrent porphyrias, administration using intravenous way for children under 5 years
* Xylocain 10 mg/ml epinephrine 0.005 mg/ml, injectable solution : Known hypersensitivity to lidocain chlorhydrate, to local amide linking anesthetic or to one of its excipients, patients affected with reccurrent porphyrias, administration using intravenous way for children under 5 years, linked to the epinephrined compound : intra vascular way, angina pectoris, ventricular rythm troubles, severe arterial hypertension, obstructive cardiomyopathy, hyper thyroidy, anesthesia with local infiltration on the extermities (fingers, penis).
* Kalinox ® (MEOPA) : Need for ventilation in pure oxygen, intracranial hypertension, alteration of consciousness, cranial trauma, pneumothorax, emphysema bubble, submarine diving accident, intestinal gas distension, gas bubble from an eye surgery under 3 months, known and non substituted B12 vitamine or folic acid deficiency, neurological disorder of recent onset and non explained.
* Person deprived from his/her freedom on a judicial or administrative decision, person under a legal protection measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2019-03-17 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Comparison of the expression of mRNA of different TRP channels between the three groups. | at the moment of the first biopsy
  Quantification of the expression of mRNA of TRP channels by RT PCR

SECONDARY OUTCOMES:
Comparison of the expression of mRNA of different TRP channels between the three groups after a loco regional cooling. | after cooling (2hours after the first biopsy)
  RT PCR
Correlation between the expression of mRNA of different TRP channels and the cutaneous blood flux between the three groups during a loco regional cooling. | after cooling (2hours after the first biopsy)
  RT PCR, laser speckle contrast imaging, infra red thermogrphy, tissue viability imaging
Correlation between the expression of mRNA of different TRP channels and the cutaneous blood flux between the three groups during a loco regional warming at 39°C and 43°C. | after warming (3 hours after the first biopsy)
  RT PCR, laser doppler
Comparison of the expression of mRNA of different TRP channels between the biopsies of an affected area (surrouding nail area) and a non-affected area (gluteal region) in the three groups. | at the moment of the biopsies
  RT PCR
Comparison of expressed micro RNA between the three groups. | at the moment of the first biopsy
  RT PCR
Comparison of the methylation states of CpG clusters found at the level of dysregulated genes. | at the moment of the first biopsy
  RT PCR
Comparison of the proportion of myo fibroblasts with or without pharmacological modulation on the TRP(s) which expression is modified in RP. | second sequence (The interval between the two sequence must not exceed 180 days)
  Immuno fluorescence with an anti-alpha smooth muscle cell antibody

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Blaise, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU of Grenoble Alpes, Grenoble, Isère, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Herrick AL. Pathogenesis of Raynaud's phenomenon. Rheumatology (Oxford). 2005 May;44(5):587-96. doi: 10.1093/rheumatology/keh552. Epub 2005 Mar 1. PMID 15741200
- [Background] Maricq HR, Carpentier PH, Weinrich MC, Keil JE, Franco A, Drouet P, Poncot OC, Maines MV. Geographic variation in the prevalence of Raynaud's phenomenon: Charleston, SC, USA, vs Tarentaise, Savoie, France. J Rheumatol. 1993 Jan;20(1):70-6. PMID 8441170
- [Background] Chifflot H, Fautrel B, Sordet C, Chatelus E, Sibilia J. Incidence and prevalence of systemic sclerosis: a systematic literature review. Semin Arthritis Rheum. 2008 Feb;37(4):223-35. doi: 10.1016/j.semarthrit.2007.05.003. Epub 2007 Aug 9. PMID 17692364
- [Background] Gabrielli A, Avvedimento EV, Krieg T. Scleroderma. N Engl J Med. 2009 May 7;360(19):1989-2003. doi: 10.1056/NEJMra0806188. No abstract available. PMID 19420368
- [Background] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Ellen Csuka M, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American college of rheumatology/European league against rheumatism collaborative initiative. Ann Rheum Dis. 2013 Nov;72(11):1747-55. doi: 10.1136/annrheumdis-2013-204424. PMID 24092682
- [Background] Steen V, Denton CP, Pope JE, Matucci-Cerinic M. Digital ulcers: overt vascular disease in systemic sclerosis. Rheumatology (Oxford). 2009 Jun;48 Suppl 3:iii19-24. doi: 10.1093/rheumatology/kep105. PMID 19487218
- [Background] Hachulla E, Clerson P, Launay D, Lambert M, Morell-Dubois S, Queyrel V, Hatron PY. Natural history of ischemic digital ulcers in systemic sclerosis: single-center retrospective longitudinal study. J Rheumatol. 2007 Dec;34(12):2423-30. Epub 2007 Nov 1. PMID 17985402
- [Background] Thompson AE, Shea B, Welch V, Fenlon D, Pope JE. Calcium-channel blockers for Raynaud's phenomenon in systemic sclerosis. Arthritis Rheum. 2001 Aug;44(8):1841-7. doi: 10.1002/1529-0131(200108)44:83.0.CO;2-8. PMID 11508437
- [Background] Roustit M, Blaise S, Allanore Y, Carpentier PH, Caglayan E, Cracowski JL. Phosphodiesterase-5 inhibitors for the treatment of secondary Raynaud's phenomenon: systematic review and meta-analysis of randomised trials. Ann Rheum Dis. 2013 Oct;72(10):1696-9. doi: 10.1136/annrheumdis-2012-202836. Epub 2013 Feb 20. PMID 23426043
- [Background] Scorza R, Caronni M, Mascagni B, Berruti V, Bazzi S, Micallef E, Arpaia G, Sardina M, Origgi L, Vanoli M. Effects of long-term cyclic iloprost therapy in systemic sclerosis with Raynaud's phenomenon. A randomized, controlled study. Clin Exp Rheumatol. 2001 Sep-Oct;19(5):503-8. PMID 11579708
- [Background] Herrick AL. Vascular function in systemic sclerosis. Curr Opin Rheumatol. 2000 Nov;12(6):527-33. doi: 10.1097/00002281-200011000-00009. PMID 11092203
- [Background] Cooke JP, Marshall JM. Mechanisms of Raynaud's disease. Vasc Med. 2005 Nov;10(4):293-307. doi: 10.1191/1358863x05vm639ra. PMID 16444858
- [Background] Toth BI, Olah A, Szollosi AG, Biro T. TRP channels in the skin. Br J Pharmacol. 2014 May;171(10):2568-81. doi: 10.1111/bph.12569. PMID 24372189
- [Background] Moran MM, McAlexander MA, Biro T, Szallasi A. Transient receptor potential channels as therapeutic targets. Nat Rev Drug Discov. 2011 Aug 1;10(8):601-20. doi: 10.1038/nrd3456. PMID 21804597
- [Background] Wong BJ, Fieger SM. Transient receptor potential vanilloid type-1 (TRPV-1) channels contribute to cutaneous thermal hyperaemia in humans. J Physiol. 2010 Nov 1;588(Pt 21):4317-26. doi: 10.1113/jphysiol.2010.195511. PMID 20807792
- [Background] Zholos A. Pharmacology of transient receptor potential melastatin channels in the vasculature. Br J Pharmacol. 2010 Apr;159(8):1559-71. doi: 10.1111/j.1476-5381.2010.00649.x. Epub 2010 Mar 5. PMID 20233227
- [Background] Wilkins BW. Bring on the heat: transient receptor potential vanilloid type-1 (TRPV-1) channels as a sensory link for local thermal hyperaemia. J Physiol. 2010 Nov 1;588(Pt 21):4065. doi: 10.1113/jphysiol.2010.199703. No abstract available. PMID 21037313
- [Background] Szabo A, Czirjak L, Sandor Z, Helyes Z, Laszlo T, Elekes K, Czompoly T, Starr A, Brain S, Szolcsanyi J, Pinter E. Investigation of sensory neurogenic components in a bleomycin-induced scleroderma model using transient receptor potential vanilloid 1 receptor- and calcitonin gene-related peptide-knockout mice. Arthritis Rheum. 2008 Jan;58(1):292-301. doi: 10.1002/art.23168. PMID 18163477
- [Background] Roustit M, Millet C, Blaise S, Dufournet B, Cracowski JL. Excellent reproducibility of laser speckle contrast imaging to assess skin microvascular reactivity. Microvasc Res. 2010 Dec;80(3):505-11. doi: 10.1016/j.mvr.2010.05.012. Epub 2010 Jun 9. PMID 20542492
- [Background] Fava A, Wung PK, Wigley FM, Hummers LK, Daya NR, Ghazarian SR, Boin F. Efficacy of Rho kinase inhibitor fasudil in secondary Raynaud's phenomenon. Arthritis Care Res (Hoboken). 2012 Jun;64(6):925-9. doi: 10.1002/acr.21622. Epub 2012 Jan 24. PMID 22275160
- [Background] Roustit M, Cracowski JL. Assessment of endothelial and neurovascular function in human skin microcirculation. Trends Pharmacol Sci. 2013 Jul;34(7):373-84. doi: 10.1016/j.tips.2013.05.007. Epub 2013 Jun 21. PMID 23791036
- [Background] Pauling JD, Shipley JA, Raper S, Watson ML, Ward SG, Harris ND, McHugh NJ. Comparison of infrared thermography and laser speckle contrast imaging for the dynamic assessment of digital microvascular function. Microvasc Res. 2012 Mar;83(2):162-7. doi: 10.1016/j.mvr.2011.06.012. Epub 2011 Jul 1. PMID 21763703
- [Background] Daly SM, Leahy MJ. 'Go with the flow ': a review of methods and advancements in blood flow imaging. J Biophotonics. 2013 Mar;6(3):217-55. doi: 10.1002/jbio.201200071. Epub 2012 Jun 18. PMID 22711377
- [Background] Johnson CD, Melanaphy D, Purse A, Stokesberry SA, Dickson P, Zholos AV. Transient receptor potential melastatin 8 channel involvement in the regulation of vascular tone. Am J Physiol Heart Circ Physiol. 2009 Jun;296(6):H1868-77. doi: 10.1152/ajpheart.01112.2008. Epub 2009 Apr 10. PMID 19363131
- [Background] Thompson AE, Pope JE. Calcium channel blockers for primary Raynaud's phenomenon: a meta-analysis. Rheumatology (Oxford). 2005 Feb;44(2):145-50. doi: 10.1093/rheumatology/keh390. Epub 2004 Nov 16. PMID 15546967